CLINICAL TRIAL: NCT04259112
Title: Effect of Pneumoperitoneum Pressure and the Extent of Neuromuscular Block on Renal Function in Patients With Diabetes Undergoing Laparoscopic Pelvic Surgery
Brief Title: Effect of Pneumoperitoneum and Neuromuscular Block on Renal Function in Diabetes Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Huang YuGuang, Dean of the Department of Anesthesiology, Peking Union Medical College Hospital
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: PUMCH-ml
Record Dates: First submitted 2020-02-02; First posted 2020-02-06 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Diabetes Mellitus; Acute Kidney Injury; Laparoscopic Surgical Procedure; Neuromuscular Blockade
MeSH Terms: conditions — Diabetes Mellitus; Acute Kidney Injury

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The patients, surgeons and the ones who collect data will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- high pressure + deep block (Experimental): Intra-abdominal pressure will be set to 12-15 mmHg during the surgery. Deep neuromuscular block will be induced by rocuronium bolus 1 mg/kg, maintained by a continuous infusion of rocuronium (0.6mg/kg/h), and titrated towards post-tetanic count (PTC) 1-2.
  Interventions: Procedure: high pressure; Drug: deep neuromuscular block
- high pressure + moderate block (Experimental): Intra-abdominal pressure will be set to 12-15 mmHg during the surgery. Moderate neuromuscular block will be induced by rocuronium bolus 0.6 mg/kg, maintained by a continuous infusion of rocuronium (0.3mg/kg/h), and titrated towards train-of-four (TOF) twitch 1-2.
  Interventions: Procedure: high pressure; Drug: moderate neuromuscular block
- low pressure + deep block (Experimental): Intra-abdominal pressure will be set to 7-10 mmHg during the surgery. Deep neuromuscular block will be induced by rocuronium bolus 1 mg/kg, maintained by a continuous infusion of rocuronium (0.6mg/kg/h), and titrated towards PTC 1-2.
  Interventions: Drug: deep neuromuscular block; Procedure: low pressure
- low pressure + moderate block (Experimental): Intra-abdominal pressure will be set to 7-10 mmHg. Moderate neuromuscular block will be induced by rocuronium bolus 0.6 mg/kg, maintained by a continuous infusion of rocuronium (0.3mg/kg/h), and titrated towards TOF twitch 1-2.
  Interventions: Drug: deep neuromuscular block; Drug: moderate neuromuscular block

INTERVENTIONS:
Procedure: high pressure — High-pressure pneumoperitoneum is defined as intra-abdominal pressure 12-15 mmHg.
  Arms: high pressure + deep block; high pressure + moderate block
Drug: deep neuromuscular block — Deep neuromuscular block is defined as PTC 1-2.
  Arms: high pressure + deep block; low pressure + deep block; low pressure + moderate block
Procedure: low pressure — Low-pressure pneumoperitoneum is defined as intra-abdominal pressure 7-10 mmHg.
  Arms: low pressure + deep block
Drug: moderate neuromuscular block — Moderate neuromuscular block is defined as TOF twitch 1-2.
  Arms: high pressure + moderate block; low pressure + moderate block

SUMMARY:
In this single center, double-blind, randomized controlled clinical trial, we will include 648 diabetes patients aged 18-70 undergoing laparoscopic pelvic tumor resection. They will be randomized to the following four groups: high-pressure pneumoperitoneum (10mmHg)+ deep neuromuscular block group, high-pressure pneumoperitoneum (15mmHg)+moderate neuromuscular block group, low-pressure pneumoperitoneum + deep neuromuscular block group and low-pressure pneumoperitoneum+moderate neuromuscular block group. Deep neuromuscular block is defined as post tetanic count (PTC) 1-2, and low neuromuscular block is defined as train-of-four (TOF) twitch 1-2. The outcomes will be indicators for acute kidney injury and surgical condition.

DETAILED DESCRIPTION:
In this single center, double-blind, randomized controlled clinical trial, we will include 648 diabetes patients aged 18-70 undergoing laparoscopic pelvic tumor resection under general anesthesia. They will be randomized to the following four groups: high-pressure pneumoperitoneum (10mmHg)+ deep neuromuscular block group, high-pressure pneumoperitoneum (15mmHg)+moderate neuromuscular block group, low-pressure pneumoperitoneum + deep neuromuscular block group and low-pressure pneumoperitoneum+moderate neuromuscular block group. Neuromuscular block will be induced by rocuronium bolus and maintained by a continuous infusion of rocuronium. Deep neuromuscular block is defined as PTC 1-2, and low neuromuscular block is defined as train-of-four TOF twitch 1-2. The primary outcome will be serum Cystatin C level, and the secondary outcomes will be serum creatine level, urinary sediment, intraoperative urine output, duration of surgery, surgical space condition and occurrence bucking and body movement.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-70;
2. American Society of Anesthesiologist physical status (ASA) II-Ⅲ;
3. Diagnosed of diabetes;
4. Undergoing elective laparoscopic pelvic tumor resection under general anesthesia;
5. Estimated duration of operation >2h;

Exclusion criteria:

1. Not willing to participate in the study or not able to sign the informed consent；
2. Diagnosed of other kidney diseases except diabetic nephropathy;
3. Severe renal insufficiency defined as serum creatine level > 2 times the upper limit of normal, or urine output < 0.5ml/kg/h, or estimated glomerular filtration rate < 60ml/h;
4. Severe liver, lung or heart dysfunction;
5. Known or suspect neuromuscular disease;
6. Use of drugs that may affect neuromuscular block monitoring;
7. Severe diabetic neuropathy or other peripheral neuropathy；
8. Known or suspect allergy to general anesthetics；
9. Family history of malignant hyperthermia；
10. Previous history of pelvic surgery.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 648 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Serum cystatin C (CysC) level | 30 minutes before pneumoperitoneum insufflation
  CysC is a sensitive indicator for early kidney injury, and can be used to estimate glomerular filtration rate (GFR).
Serum cystatin C (CysC) level | 30 minutes after pneumoperitoneum deflatation
  CysC is a sensitive indicator for early kidney injury, and can be used to estimate glomerular filtration rate (GFR).
Serum cystatin C (CysC) level | Postoperative 24 hours
  CysC is a sensitive indicator for early kidney injury, and can be used to estimate glomerular filtration rate (GFR).

SECONDARY OUTCOMES:
Serum creatine level | 30 minutes before pneumoperitoneum insufflation
  Creatine is also an indicator for kidney injury
Serum creatine level | 30 minutes after pneumoperitoneum deflatation
  Creatine is also an indicator for kidney injury
Serum creatine level | Postoperative 24 hours
  Creatine is also an indicator for kidney injury
The volume of intraoperative urine output | At the end of the surgery
  A urine tube will be inserted just before the surgery, so the urine can be drained into a bag. The volume of urine in the bag at the end of the surgery will be the volume of intraoperative urine output.
The presence of isomorphic or dysmorphic erythrocyte in urinary sediment | Postoperative day 1
  Erythrocyte in urinary sediment is also an indicator of renal injury.
Duration of surgery | Intraoperative
  Duration of surgery is an indicator for procedure difficulty
Leiden-surgical rating scale | The moment when trocars are introduced into pelvic cavity, and then every 15 minutes till the end of surgery.
  We will use Leiden surgical rating scale (Martini et al.) to assess surgical condition. It is a 5-point scale, the minimum and maximum values are 1 and 5, respectively. Higher score indicates better surgical condition.
The number of bucking and body movement during the surgery | Intraoperative
  The occurrence of bucking or body movement is an indicator for the sufficiency of muscle relaxant.
Renal tissue oxygen saturation | Intraoperative
  Renal oxygen saturation is an indicator for renal tissue oxygenation.

CONTACTS AND LOCATIONS:
Overall Officials: Yuguang Huang, M.D., Principal Investigator — Peking Union Medical College Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xu X, Gong Y, Zhang Y, Lang J, Huang Y. Effect of pneumoperitoneum pressure and the depth of neuromuscular block on renal function in patients with diabetes undergoing laparoscopic pelvic surgery: study protocol for a double-blinded 2 x 2 factorial randomized controlled trial. Trials. 2020 Jun 29;21(1):585. doi: 10.1186/s13063-020-04477-x. PMID 32600358